CLINICAL TRIAL: NCT05881161
Title: Bridging the Adherence Gap in Internet Interventions: A Randomized Controlled Trial Study Protocol Investigating Context-Specific Self-Efficacy
Brief Title: Bridging the Adherence Gap in Internet Interventions: A Randomized Controlled Trial Protocol
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Sciences and Humanities, Warsaw (Other)
Collaborators: Stockholm University (Other)
Responsible Party: Principal Investigator, Ewelina Smoktunowicz, Principal Investigator; Head of StresLab Research Centre, University of Social Sciences and Humanities, Warsaw
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Adherence
Record Dates: First submitted 2023-05-18; First posted 2023-05-31 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Adherence, Treatment; Job Stress
Keywords: Job Stress; Adherence; Work engagement; Self-efficacy
MeSH Terms: conditions — Treatment Adherence and Compliance; Occupational Stress

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not be informed about condition allocation. Both groups will undergo the same internet intervention (Med-Stress Student) but the experimental group will complete additional procedure at the start of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adherence self-efficacy-enhancing exercise followed by internet intervention (Med-Stress Student) (Experimental)
  Interventions: Behavioral: Adherence self-efficacy-enhancing exercise; Behavioral: Med-Stress Student
- Internet intervention (Med-Stress Student) (Active Comparator)
  Interventions: Behavioral: Med-Stress Student

INTERVENTIONS:
Behavioral: Adherence self-efficacy-enhancing exercise — This exercise aims to increase self-efficacy to adhere to an internet intervention. It consists of a video and two text-based tasks. The contents are grounded in Social-Cognitive Theory.
  Arms: Adherence self-efficacy-enhancing exercise followed by internet intervention (Med-Stress Student)
Behavioral: Med-Stress Student — Med-Stress Student is an intervention that spans over 4 weeks and aims to enhance resources to cope with job stress and promote well-being in medical students.

SUMMARY:
Low adherence in self-guided internet interventions might lead to worse outcomes. This randomized controlled trial aims to test whether adherence can be improved if self-efficacy regarding adherence to internet interventions is boosted before the intervention starts. It is expected that enhancing this specific type of self-efficacy will increase people's adherence and help them fully benefit from the intervention, namely experience lower job stress and higher work engagement.

DETAILED DESCRIPTION:
Low adherence can lead to poor outcomes in self-guided (i.e., self-administered) internet interventions that is psychological programs designed to improve mental health. One modifiable personal factor that may improve adherence is context-specific self-efficacy. In this two-arm randomized controlled trial, participants (medical students, N = 720) will undergo an internet intervention called Med-Stress Student designed to enhance resources such as self-efficacy to cope with stress and perceived social support. In the experimental group, Med-Stress Student will be preceded by an exercise designed to boost self-efficacy to adhere to this internet intervention. In the control condition, participants will only access Med-Stress Student. Conditions will be compared on adherence as well as on the intervention outcomes (i.e., job stress and work engagement) at posttest, and at six-month, and one-year follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* must be at least 18 years old
* must be a medical student or intern who already has direct contact with patients

There are no criteria for exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 952 (Estimated)
Dates: Start 2025-01-08 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Adherence | Change from baseline: 4 weeks (posttest)
  Objective adherence will be based on quantifiable metrics, specifically the absolute number and percentage of completed exercises within the program. Subjective adherence will be evaluated with the following question that participants will respond to after each weekly set of exercises: "In your opinion, how accurately have you completed all tasks: have you followed the instructions, reflected on the questions, and responded to them exhaustively?".

SECONDARY OUTCOMES:
Job Stress (Perceived Stress Scale; PSS-4) | Change from baseline: 4 weeks (posttest)
  The brief version of the scale consists of four items, rated on a scale ranging from 0 (never) to 4 (very often). It will be applied to measure job stress, with a higher total score indicating a heightened level of stress perception. The questionnaire's instructions have been modified to align with the occupational context.
Job Stress (Perceived Stress Scale; PSS-4) | Change from baseline: 1-year follow-up
  The brief version of the scale consists of four items, rated on a scale ranging from 0 (never) to 4 (very often). It will be applied to measure job stress, with a higher total score indicating a heightened level of stress perception. The questionnaire's instructions have been modified to align with the occupational context.
Job Stress (Perceived Stress Scale; PSS-4) | Change from baseline: 6-month follow-up
  The brief version of the scale consists of four items, rated on a scale ranging from 0 (never) to 4 (very often). It will be applied to measure job stress, with a higher total score indicating a heightened level of stress perception. The questionnaire's instructions have been modified to align with the occupational context.
Work Engagement (Utrecht Work Engagement Scale; UWES-9) | Change from baseline: 6-month follow-up
  A 9-item variant of the scale will be used to assess work engagement. The response range varies between 0 (never) and 6 (always), with a higher total score signifying greater work engagement.
Work Engagement (Utrecht Work Engagement Scale; UWES-9) | Change from baseline: 1-year follow-up
  A 9-item variant of the scale will be used to assess work engagement. The response range varies between 0 (never) and 6 (always), with a higher total score signifying greater work engagement.
Work Engagement (Utrecht Work Engagement Scale; UWES-9) | Change from baseline: 4 weeks (posttest)
  A 9-item scale will be used to assess work engagement. The response range varies between 0 (never) to 6 (always), with a higher total score indicating a higher work engagement.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Karyotaki E, Kleiboer A, Smit F, Turner DT, Pastor AM, Andersson G, Berger T, Botella C, Breton JM, Carlbring P, Christensen H, de Graaf E, Griffiths K, Donker T, Farrer L, Huibers MJ, Lenndin J, Mackinnon A, Meyer B, Moritz S, Riper H, Spek V, Vernmark K, Cuijpers P. Predictors of treatment dropout in self-guided web-based interventions for depression: an 'individual patient data' meta-analysis. Psychol Med. 2015 Oct;45(13):2717-26. doi: 10.1017/S0033291715000665. Epub 2015 Apr 17. PMID 25881626
- [Background] Smoktunowicz E, Lesnierowska M, Carlbring P, Andersson G, Cieslak R. Resource-Based Internet Intervention (Med-Stress) to Improve Well-Being Among Medical Professionals: Randomized Controlled Trial. J Med Internet Res. 2021 Jan 11;23(1):e21445. doi: 10.2196/21445. PMID 33427674